CLINICAL TRIAL: NCT05101824
Title: Bony M - Stereotactic Ablative Radiotherapy (SABR) of Bony Metastases in Patients With Oligometastatic Disease - A Phase II Study
Brief Title: Bony M - Stereotactic Ablative Radiotherapy (SABR) of Bony Metastases in Patients With Oligometastatic Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gitte Fredberg Persson MD PhD (Other)
Responsible Party: Sponsor-Investigator, Gitte Fredberg Persson MD PhD, Associate professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-19039071
Record Dates: First submitted 2021-03-25; First posted 2021-11-01 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Oligometastatic Disease; Bone Metastases; Stereotactic Body Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single arm, multicenter, phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): All recruited patients are treated with SABR.
  Interventions: Radiation: SABR

INTERVENTIONS:
Radiation: SABR — Two fractionation regimes are available (37.5 Gy in 3 fractions and 30.0 Gy in 3 fractions)

SUMMARY:
This is a prospective, investigator-initiated, phase II, multicentre-study, investigating the efficacy and toxicity of definitive SABR of osseous oligometastases, when pragmatically introduced into a daily clinical setting.

DETAILED DESCRIPTION:
Patients with a histology or cytology proven non-hematological cancer and at least one lesion in the bones are eligible.

Patients with de novo- and induced oligometastatic disease, as well as patients with oligo-recurrence or oligo-progression disease can be included. A total of 67 patients will be enrolled.

The overall aim is to document long time follow-up in respect to local control rate, OS, PFS, rate of symptomatic skeletal event at the irradiated site(s), time to progression outside the radiation field at 1-, 2- and 5-years and acute/ late toxicities.

The primary endpoint is the rate of local control 1-year post SABR. Patients will have a CT scan and a clinical evaluation every 3 month after SABR according to the standard clinical follow-up program.

During the 1 year follow-up we also perform pain assessment (using the Numeric Pain Rating Scale), report the analgesic consumption and Quality of life (QoL) measured with EQ-5D-5L.

Two dose levels are offered with either 37.5 gy in 3 fractions or 30 gy in 3 fractions, prescribed to the GTV.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology proven non-haematological cancer.
* At least one lesion in the bones is required.
* ECOG performance status ≤ 2.
* ≥ 18 years old.
* Life expectancy > 6 months.
* GTV diameter ≤ 5 cm.
* In case of de novo OMD and OMD recurrence a maximum of 5 targets (including the primary tumour) in a maximum of 3 organ sites are allowed.
* In case of OPD * and induced OMD*2 only 3 metastases (including the primary tumour) are allowed.
* The metastatic lesion(s) must be visible on a CT- or MR- scan and suitable for treatment with SABR.
* All metastatic sites are treated or planned for ablative therapy (including surgery) - for OPD only the sites in progression is required to fulfil this criterion. • A baseline scan within 28 days of inclusion (CT or PET- CT).
* For spine/paraspinal targets, an MR scan is mandatory, if epidural growth cannot be precluded on the baseline CT scan.
* No curative intended treatment option available.
* An ablative strategy should be deemed clinically relevant and is at the discretion of the treating physician to decide.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patient cannot tolerate physical set up required for SABR.
* Uncontrolled intercurrent illness.
* Pregnancy.
* Bilsky score ≥ 1b. If the patient is treated with surgery, a pre-operative Bilsky score ≥ 1b is an exclusion criterion as well. See appendix A for Bilsky score.
* Presence of myelopathy from the target area.
* Candidate for surgical treatment (determined by the institutions clinical oncologist, neurosurgeon or orthopaedic surgeon).
* For spine/paraspinal lesions where epidural growth cannot be precluded on the baseline CT scan: patients for whom an MR scan is contraindicated.
* Mechanical instability and/or fracture risk *3.
* For spine disease, involvement of ≥ three contiguous vertebrae.
* Uncontrolled disease in respect to malignant pleural effusion, ascites, lymphangitic carcinomatosis, pleural carcinomatosis or peritoneal carcinomatosis.
* Patients with uncontrolled brain metastases.
* If the patient has received previous radiotherapy, the combined dose at the radiation site must not exceed the dose constraints according to Appendix B. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
local control rate (LC) at 1-year post SABR | 1-year post SABR
  Response evaluation is based on the interpretation of a experienced onco-radiologist and modifications from the MDACC response criteria's.

SECONDARY OUTCOMES:
Rate of Symptomatic Skeletal Event (SSE) at the irradiated site(s) | 3-, 6-, 12- and 24-months post SBRT
  Symptomatic Skeletal Event (SSE) of the irradiated site is defined as a radiographically verification of fracture (vertebral or non-vertebral, pathological or non-pathological), within or adjacent to the PTV of the irradiated site. The fracture must co-exist with one of the
Pain, change from baseline evaluated by "Numeric Pain Rating Scale (NPRS)" | Measured at 2-, 12-, 24-, 36- and 52-weeks post SBRT
  Response categories is based on patient reported pain scores (NPRS). The 11- 9 Protocol version 1.1, 01052020. Stereotactic ablative radiotherapy (SABR) of bony metastases in patients with oligometastatic disease - A phase II study point NPRS ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
NCI CTCAE ≥ grade 3 toxicity | Measured at 2-, 12-weeks post SBRT
  Cummulated fraction of patients, who encounter one or more ≥ grade 3 NCI CTCAE toxicity within the first 3-months after SBRT.
NCI CTCAE ≥ grade 3 late toxicity | Measured at 3-, 6-, 12- and 24-months post SBRT
  Cummulated fraction of patients, who encounter one or more ≥ grade 3 NCI CTCAE toxicity from 3-months and onward after SBRT including patients who have unresolved early toxicity (encontered within the first 3-months), that is not resolved at the 24-weeks follow-up.
Local progression free survival | continuous within 2-years post SBRT
  Local progression free survival is defined as time from inclusion until progression of the irradiated lesion. Patients are not censored from analysis in case of new lesions outside the irradiated volume. The irradiated volume is defined as, within or adjacent to the PTV. Local progression free survival is reported as a continuos variable.
Progression-free survival (PFS) | Continuous and at 3-, 6-, 12- and 24-months post SBRT
  Progression-free survival is defined as time from inclusion until disease progression or death following symptoms/interventions: progression in pain (according to definition in section 3.5), development of neurological symptoms/ symptomatic spinal cord compression or a need for surgical intervention/ reirradiation. It should be concluded from the treating physician that the symptom/intervention is a result of the fracture. Vertebral fractures include end plate-only fractures. Analysis is done at a lesion level, lesion by lesion. Patients with a pathological fracture before the radiation therapy, will not be included for analysis
Time to progression (TTP) outside the radiation field | Continuous and at 3-, 6-, 12- and 24-months post SBRT
  Time to progression outside the radiation field is defined, as the time from inclusion until progression outside the radiation field, determined by a CT -, MR -, or PET-CT - scan. Outside the radiation field is defined as outside and not adjacent to the PTV.
Overall survival (OS) | continuous till 2-year post SABR
  OS is defined as time from inclusion until death from any cause
Quality of life (QoL) measured with EQ-5D-5L. | at 3-, 6-, 12- and 24-months post SBRT
  Change from baseline in mobility using the 5-level system in EQ-5D-5L
Quality of life (QoL) measured with EQ-5D-5L. | at 3-, 6-, 12- and 24-months post SBRT
  Change from baseline in self-care score using the 5-level system in EQ-5D-5L
Quality of life (QoL) measured with EQ-5D-5L. | at 3-, 6-, 12- and 24-months post SBRT
  Change from baseline in usual activities score using the 5-level system in EQ-5D-5L.
Quality of life (QoL) measured with EQ-5D-5L. | at 3-, 6-, 12- and 24-months post SBRT
  Change from baseline in pain/discomfort score using the 5-level system in EQ-5D-5L.
Quality of life (QoL) measured with EQ-5D-5L. | at 3-, 6-, 12- and 24-months post SBRT
  Change from baseline in anxiety/depression score using the 5-level system in EQ-5D-5L.
Quality of life (QoL) measured with EQ-5D-5L. | at 3-, 6-, 12- and 24-months post SBRT
  Change from baseline in self assessed EQ visual analogue scale in EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Persson, Principal Investigator — Hospital of Herlev and Gentifte
Locations (6):
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- Norway (2):
  - Ålesund sjukehus, Ålesund
  - St Olavs Universitetssykehus,, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spindler NJ, Felter MVO, Hansen O, Nielsen TB, Suppli MH, Josipovic M, Poulsen LO, Rahma-Petersen F, Sand HMB, Abramova TM, Johansen M, Kornerup JS, Alsaker MD, Eefsen RL, Serup-Hansen E, Andersen MB, Geertsen P, Vogelius IR, Behrens CP, Persson GF. Stereotactic Ablative Radiation Therapy of Bone Metastases in an Oligometastatic Setting: One-Year Follow-Up of the BONY-M Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2025 Jul 24:S0360-3016(25)06023-7. doi: 10.1016/j.ijrobp.2025.07.1419. Online ahead of print. PMID 40714134

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT05101824/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT05101824/SAP_001.pdf